CLINICAL TRIAL: NCT04393571
Title: The Utility of Mobile Based Patient Reported Outcome Measures(PROMS) in Patients With Acetabular Fractures: A Randomized Controlled Trial.
Brief Title: The Utility of Mobile Based Patient Reported Outcome Measures in Patients With Acetabular Fractures: A Randomized Controlled Trial.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Collaborators: AO Trauma (Unknown)
Responsible Party: Principal Investigator, Mohammed Kamal Abdelnasser, clinical professor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TUOMBPROMSIPWAFARCT
Record Dates: First submitted 2020-05-03; First posted 2020-05-19 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Acetabular Fracture; PROMs; Mobile Phone Use
MeSH Terms: conditions — Cell Phone Use

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional follow up patients (Experimental)
  Interventions: Other: Mobile application
- Mobile app follow up patients (Experimental)
  Interventions: Other: Mobile application

INTERVENTIONS:
Other: Mobile application — telemedicine is used to overcome distance when patients must travel to receive specialized care. We depend on the available, widely used smartphones via a mobile application to conduct follow up data as regard to patient quality of life and comparing this to conventional follow up visits and whether it help to obtain a complete follow up data

SUMMARY:
Acetabular fractures are articular fractures involving the hip joint that needs anatomical reduction and a strict long follow up after fixation.

DETAILED DESCRIPTION:
The percentage of patients with lost follow up is significantly high. Previously all other studies mainly focused on the radiographic outcome after acetabular fractures and rarely on patient reported functional outcomes and quality of life. The use of patient-reported outcome measures (PROMs) is increasing and may lead to modifications of treatment. Recent technologic advances, namely smartphones, capable of measuring outcomes after acetabular fractures are now very important in quantifying value-based care. This was previously accomplished through office assessments and surveys with variable follow-up but this strategy lacks continuous and complete data. Studies show that these remote modes of follow-up are safe and that patients are as equally satisfied with them as they are with in-person follow- up care

ELIGIBILITY:
Inclusion Criteria:

* all patients older than 18 years old who will have surgery for an acetabular fracture at assiut university hospitals from 1/10/2020 to 30/9/2022.

Exclusion Criteria:

* patients younger than 18 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2022-10-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
the percentage of missed follow up data in both groups at 12 months postoperatively | at least one year follow up
  through assessing the patient-reported outcome measures (PROMS) after surgery for a fracture of the acetabulum in assiut university hospital using the Arabic validated form of the 36-Item Short Form Health Survey (SF-36).

SECONDARY OUTCOMES:
the ability of the mobile application to rapidly detect the occurrence of serious postoperative complication. | at least one year follow up
  to record the ability of the mobile application to rapidly detect the occurrence of serious postoperative complication as infection and DVT and notify us by this complication by means of the Red Flag signs which will be added to the application.

IPD SHARING:
Plan to Share IPD: Undecided